CLINICAL TRIAL: NCT04277689
Title: Deep Neural Network Approaches for Closed-Loop Deep Brain Stimulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert Mark Richardson, Director of Functional Neurosurgery at MGH, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019P003874
Record Dates: First submitted 2020-01-08; First posted 2020-02-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain signal data collection (Experimental): Collection of brain data during deep brain stimulation
  Interventions: Procedure: Brain signal data collection

INTERVENTIONS:
Procedure: Brain signal data collection — Collection of speech related electrophysiological data at the time of DBS.

SUMMARY:
In this research study the researchers want to learn more about brain activity related to speech perception and production in patients with Parkinson's Disease who are undergoing deep brain stimulation (DBS).

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is the gold-standard treatment for patients with medication resistant motor complications of Parkinson's disease (PD) and provides the only opportunity to record and stimulate in the human basal ganglia. Most recently, the concurrent use of research electrocorticography (ECoG) during DBS surgery, including pioneering work from Pittsburgh, has further enabled basic neuroscience investigation of human cortical-subcortical network dynamics. The discovery that aberrant synchronization of rhythmic neuronal activity recorded in PD patients is suppressed by DBS has advanced the concept that measures associated with pathological activity may be used as biomarkers to control the delivery of DBS therapy. Pilot studies of aDBS in PD have reported promising clinical results from triggering DBS stimulation when the signal recorded from the DBS electrode showed a high level of oscillatory power in the beta frequency range (13 - 35 Hz). That approach, however, has important limitations. Most importantly, beta power recorded from the DBS lead is suppressed by movement including PD tremor, its detection is highly dependent on lead location and the recording montage needed to record during stimulation is incompatible with directional current steering, a recent innovation employing segmented stimulation contacts. The inherent complexity of the increased parameter space through DBS innovations also overwhelms standard programming techniques. Finally, use of additional biomarker signals (e.g., recorded from cortex) is likely to improve the ability to adaptively control DBS for disorders marked by complex multidimensional symptomatologies such as PD. The current proposal will establish methods for overcoming these limitations by developing techniques for multi-feature classification from ECoG recordings, using advanced machine learning algorithms.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled for DBS implantation, as determined by the clinical multidisciplinary movement disorders board with definitive diagnosis of Parkinson's disease
2. Subjects able to provide informed consent and comply with task instructions.
3. Subjects 18-85 years old

Exclusion Criteria:

1. Non-English-speaking subjects

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The number of subjects providing interpretable electrophysiological data during DBS surgery | Duration of single DBS surgery
  The number of subjects providing interpretable electrophysiological data during DBS surgery

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Richardson, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No